CLINICAL TRIAL: NCT01167868
Title: A Phase I, Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Assess the Safety, Tolerability and Pharmacokinetics of Oral Fostamatinib Disodium in Healthy Japanese and White Subjects After Single and Multiple Ascending Doses
Brief Title: A Study to Assess the Safety, Tolerability, and Blood and Urine Drug Levels of Fostamatinib Disodium (FosD) in Healthy Japanese and White Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D4300C00007
Record Dates: First submitted 2010-07-19; First posted 2010-07-22 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Healthy
Keywords: fostamatinib disodium; FosD; Japanese; Healthy volunteers; Phase 1; Single and Multiple Ascending Dose Study; Healthy Japanese volunteers; Healthy White volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- FosD (Experimental): Four sequential cohorts of Japanese subjects are planned with doses ranging from 50mg once daily to a maximum of 200mg twice daily. One cohort of White subjects is also planned to receive the same dose regimen as the third dose level in Japanese subjects
  Interventions: Drug: FosD
- Placebo (Placebo Comparator): Placebo given (2 subjects in each cohort)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FosD — oral tablet
  Arms: FosD
Drug: Placebo — oral tablet
  Arms: Placebo

SUMMARY:
This is a single and multiple ascending dose study in healthy male and female (of non-child bearing potential) Japanese and White volunteers, to assess the safety, tolerability, and blood and urine drug levels of FosD. FosD is being developed for the treatment of rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female (of non-childbearing potential) Japanese subjects and White subjects (origins in Europe, the Middle East, or North Africa)
* Body mass index (BMI) between 17 and 27 kg/m2 and weigh at least 45 kg and no more than 100 kg

Exclusion Criteria:

* History or presence of respiratory, GI, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders
* Any clinically significant illness, acute infection, known inflammatory process, medical/surgical procedure or trauma within 4 weeks of the first administration of investigational product
* Smoking in excess of 5 cigarettes per day or equivalent within 30 days of Day 1
* Use of prescription or over-the-counter drugs within 2 weeks of first administration of investigational product

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2010-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To investigate safety and tolerability: adverse event monitoring, vital signs, physical examinations, clinical laboratory tests, 12 lead ECG, digital ECG, telemetry. | Prior to treatment, during treatment, and a follow-up visit, a total of up to 20 days

SECONDARY OUTCOMES:
To determine plasma PK parameters (including but not limited to: AUC, tmax, Cmax, terminal elimination half life (t1/2) and accumulation ratio (Rac)) of FosD. | Plasma sampling for 72 hours following both the single dose and after 7 days repeated dosing.
To determine urine PK parameters (including but not limited to: amount excreted (Ae) and renal clearance (CLr)) of FosD. | Urine sampling for upto 48 hours following both the single dose and after 7 days repeated dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Layton, MD, Study Director — AstraZeneca; Mark Yen, MD, Principal Investigator — PAREXEL Early Phase/California Clinical Trials Medical Group
Locations (1):
- Research Site, Glendale, California, United States